CLINICAL TRIAL: NCT06855134
Title: Randomized Comparison of Treatment Guided by Comprehensive Genome and Transcriptome Analysis Versus Standard of Care in Patients with Advanced Rare Cancers (RATIONALE)
Brief Title: Treatment Guided by Comprehensive Genome and Transcriptome Analysis Versus Standard of Care in Advanced Rare Cancers
Acronym: RATIONALE
Status: Not yet recruiting | Type: Observational
Sponsor: German Cancer Research Center (Other)
Collaborators: NCT Berlin: Charité- Universitätsmedizin Berlin (Unknown); NCT Dresden: University Hospital Dresden (Unknown); NCT Heidelberg: University Hospital Heidelberg (Unknown); NCT WERA: University Hospital Würzburg, University Hospital Erlangen, University Hospital Regensburg, University Hospital Augsburg (Unknown); NCT West: University Hospital Cologne, University Hospital Essen (Unknown); NCT Southwest: University Hospital Tübingen, Robert-Bosch-Hospital Stuttgart, University Hospital Ulm (Unknown)
Responsible Party: Sponsor
Other Study IDs: TMO-2501; TMO 2501 (Other: German Cancer Research Center)
Record Dates: First submitted 2025-02-28; First posted 2025-03-03 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Rare Cancer
Keywords: Molecular tumor board; molecularly informed treatment recommendation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 48 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- MPI-arm: an immediate molecular profile-informed treatment arm (MPI arm)
- MPP-arm: standard treatment arm with molecular profile-informed treatment upon progression or intolerable toxicity after standard therapy

SUMMARY:
Rare cancers, defined by an incidence of fewer than 6 cases per 100,000 persons per year, constitute nearly 25% of adult malignancies. They are associated with poor patient outcomes due to incomplete biological understanding and inadequate representation in clinical trials. To address this gap, the DKFZ/NCT/DKTK MASTER (Molecularly Aided Stratification for Tumor Eradication Research) program, developed by NCT and DKFZ, integrates whole-genome/exome sequencing (WGS/WES), RNA sequencing (RNA-seq), and genome-wide DNA methylation profiling to inform clinical decision-making in patients with advanced rare cancers. This approach has demonstrated significant improvements in overall response rates (ORR) in 24% and disease control rates (DCR) in 55% of cases, with a progression-free survival (PFS) ratio greater than 1.3 in 36% of patients.

The randomized, multi-basket, phase II, Italian multicenter ROME study conducted among pretreated patients with metastatic cancer, demonstrated that targeted therapy guided by comprehensive genomic profiling and molecular tumor board (MTB) recommendations significantly improved overall response rate and progression-free survival. Additionally, the study revealed a substantial long-term PFS benefit extending to 12 months and beyond. Although the toxicity profiles differed between the targeted therapy and standard-of-care groups, the incidence of adverse events was comparable. These findings, reported at the ESMO Congress 2024, emphasize the pivotal role of MTBs in advancing precision oncology through a tumor agnostic, molecularly guided therapeutic approach.

The objective of the randomized, multicentric, diagnostic RATIONALE trial is to evaluate the efficacy of molecularly guided treatment versus standard treatment in patients with rare cancers by comparing progression-free survival (PFS) between the two arms: an immediate molecular profile-informed treatment arm (MPI arm) and a standard treatment arm with molecular profile-informed treatment upon progression or intolerable toxicity after standard therapy (MPP arm).

Patients with rare epithelial and mesenchymal neoplasms are evenly randomized in a 1:1 ratio to either the MPl arm or MPP arm. Comprehensive molecular profiling includes WGS and RNA-seq for both arms. A multidisciplinary MTB evaluates these molecular profiles and provides clinically relevant management recommendations, including diagnostic reevaluation, genetic counseling, and molecularly informed treatment options. Recommendations may include matching patients to molecularly stratified clinical trials or - if no suitable clinical trials can be identified - coordinated applications will be provided for off-label use in routine clinical care. The primary efficacy endpoint is progression-free survival (PFS), whereas secondary endpoints are overall survival (OS), overall response rate (ORR), disease control rate (DCR) after three and six months, and patient-reported outcomes (PROs).

Based on data from the MASTER cohort, it is anticipated a median PFS of three months with treatment selected by the physician's discretion. Drawing on findings from the CRAFT trial (ClinicalTrials.gov: NCT04551521), MTB-guided treatment is expected to positively impact the primary endpoint with a hazard ratio (HR) ranging from 0.4 to 0.6. Assuming 30% implementation rate of MTB recommendations, a sample size of 756 eligible patients will be required to demonstrate a significant improvement in PFS with immediate MTB guided treatment, yielding an HR of 0.5 for the MPI arm and overall study HR of 0.7862. The calculation is based on a type 1 error of 5% and a statistical power of 90%. Considering a conservative estimate that that 20% of patients will not be evaluable, the total rounded required sample size is 946 patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18years, no upper age limit
* Patients with locally advanced and/or metastatic rare epithelial or mesenchymal cancer (equal numbers of patients) without curative treatment option
* Progressive disease or expected progression of the disease estimated by clinical parameters, suitable biomarkers, and other (e.g. radiographic) methods * At least one measurable lesion that has been accurately assessed by computed tomography (CT) or magnetic resonance imaging (MRI) at baseline and is amenable to repeat evaluation in MRI/CT images
* Patients must have received at least one standard therapy for advanced disease according to current guidelines or consensus recommendations or have no standard therapy available
* Possibility to perform fresh tumor biopsy according to local SOPs or Availability of fresh frozen tumor samples with sufficient tumor cell content collected within 3 months prior to enrolment
* ECOG PS ≤ 2.
* Ability of patient to understand character and consequences of the clinical trial
* Patient must be willing and able to undergo subsequent treatment (e.g. in a clinical trial) with molecularly guided therapy according to the MTB recommendation
* Availability of complete information about all medical treatment given before study participation, i.e. remission status before start of treatment, dosage and timing of drugs applied, remission status and date of progression after treatment

Exclusion Criteria:

* Dementia or significant cognitive impairment
* Epilepsy requiring pharmacologic treatment
* Prior allogeneic bone marrow or solid organ transplantation
* Hematological malignancies and primary brain tumors.
* Prior comprehensive molecular profiling by WGS, WES, RNA-Seq, or large targeted panels.
* Patients with symptomatic or uncontrolled brain metastases and patients with symptomatic or uncontrolled spinal cord compression. Patients with previously treated brain metastases are eligible, provided that the patient has neither experienced a seizure nor had a clinically significant change in neurological status within the three months prior to enrollment. All patients with previously treated brain metastases must be clinically stable for at least 1 month after completion of treatment and off steroid treatment for one month, both prior to study enrollment.
* Malignancy other than study indication within the last 5 years except: curatively treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), Stage 1, grade 1 endometrial carcinoma, low-risk prostate cancer, or other malignancies curatively treated with no evidence of disease for ≥5 years.
* History of intracranial hemorrhage or spinal cord haemorrhage; no ongoing requirement for dexamethasone for CNS disease; patients on a stable dose of anticonvulsants are permitted
* Known uncontrolled or significant cardiovascular disease, including any of the following:
* History of heart failure NYHA class 3 or 4
* History of uncontrolled angina pectoris, arrhythmias, or myocardial infarction within 12 months prior to screening.
* History of liver cirrhosis
* Neurologic or psychiatric disorder interfering with ability of giving informed consent.
* Known or suspected active alcohol or drug abuse.
* Patients with inability to receive oral medications.
* Failure to provide consent for the registration, storage, and processing of individual disease characteristics and clinical course, as well as for informing the primary care physician about the participant's involvement in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced and/or metastatic rare epithelial or mesenchymal cancer (equal numbers of patients) without curative treatment option
Sampling Method: Probability Sample
Enrollment: 946 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2029-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 48 months
  Progression free survival (PFS) measured from (i) start of the genomics-guided treatment or (ii) standard-of-care treatment started after randomization until radiographic disease progression or death, whatever occurs first. Patients alive and progression-free are censored at last tumor measurement according to radiographic and disease-specific assessment. For patients undergoing active tumor therapy before randomization (bridging treatment), PFS is measured from (i) start of the genomics-guided treatment or (ii) standard-of-care treatment started following the bridging treatment until radiographic disease progression or death,
  whatever occurs first.

SECONDARY OUTCOMES:
Overall Survival | 48 months
  Overall Survival (OS), the time from randomization until death from any cause. Patients without event are censored on the last date of follow-up.
R-progression free survival | 48months
  rPFS, defined as the time from randomization to time of progression of the disease or death from any cause, whatever occurs first.
MR-progression free survival | 48 months
  mrPFS, defined as the time from release of MTB report to time of progression of the disease or death from any cause, whatever occurs first.
Paired Progression Free Survival | 48 months
  Paired Progression Free Survival (PFS ratio) observed with genomic guided treatment (PFS2) and Progression Free Survival observed directly before genomics-guided treatment (PFS1)
Overall response rate | 6 months
  Overall Response rate (ORR), defined as the proportion of patients with complete response (CR) or partial response (PR) as assessed per RECIST v1.1 at 3 and 6 months after start of the recommended therapy is analyzed.
Disease control rate | 6 months
  Disease Control Rate (DCR), defined as the proportion of patients with CR, PR or stable disease (SD) as assessed per RECIST v1.1. DCR at 3 and 6 months after start of the recommended therapy is analyzed.
Health related quality of live | 6 months
  HRQoL, measured using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) as presented in patient-reported outcomes.
molecular tumor board recommendation rate | 3 months
  MTB recommendation rate, defined as the proportion of patients who receive therapeutic recommendations in the MTB

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Fröhling, MD, Principal Investigator — German Cancer Research Center; Hanno Glimm, MD, Principal Investigator — Technische Universität Dresden; Richard F Schlenk, MD, Principal Investigator — University Hospital Heidelberg

IPD SHARING:
Plan to Share IPD: Yes
IPD are shared within the German NCT-network and the German Cancer Research Center
Supporting Information: Study Protocol, ICF
Time Frame: April 2023 - undefined
Access Criteria: Researches within the German NCT-network and the German Cancer Research Center. Access is possible via a central secondary use database